CLINICAL TRIAL: NCT06274411
Title: Standby Cannulated ECMO Versus Prophylactic ECMO In Patients Undergoing High-Risk Percutaneous Coronary Intervention
Brief Title: Standby Cannulated ECMO for High-Risk Percutaneous Coronary Intervention
Acronym: ECMO-READY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Wuhan Asia Heart Hospital (Other); The First Hospital of Jilin University (Other); First Affiliated Hospital of Harbin Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); The First Affiliated Hospital of Lanzhou Medical University (Unknown); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other); First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Xiaotong Hou, Professor, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KS2024014
Record Dates: First submitted 2023-12-24; First posted 2024-02-23 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: ECMO; High-risk PCI
Keywords: ECMO; PCI

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standby cannulated ECMO (Experimental): For standby cannulated ECMO procedures, femoral cannulas are inserted either by percutaneous approach or surgical approach. The primed circuit is connected to the inserted ECMO cannulas, clamps are kept on circuit, and ECMO is on standby during PCI. When PCI cause hemodynamic instability, clamps on circuit are removed, and VA-ECMO is initiated to maintain maintain adequate systemic pressure and perfusion.
  Interventions: Procedure: Standby cannulated ECMO
- Prophylactic ECMO (Active Comparator): Prophylactic ECMO procedures are performed in the catheterization laboratory before PCI. Femoral cannulas are inserted either by percutaneous approach or surgical approach. Following cannula placement, VA-ECMO is initiated to maintain adequate systemic pressure and perfusion during PCI.
  Interventions: Procedure: Prophylactic ECMO

INTERVENTIONS:
Procedure: Standby cannulated ECMO — Femoral cannulas are inserted and connected to the primed circuit. Clamps are kept on circuit, and ECMO is on standby during PCI. ECMO is initiated if needed.
  Arms: Standby cannulated ECMO
Procedure: Prophylactic ECMO — Prophylactic ECMO procedures are performed in the catheterization laboratory before PCI.
  Arms: Prophylactic ECMO

SUMMARY:
The goal of this multicenter, randomized trial is to compare standby cannulated ECMO versus prophylactic ECMO in patients undergoing high-risk percutaneous coronary intervention (PCI). The main question it aims to answer is :

• If standby cannulated ECMO as compared with prophylactic ECMO will improve the outcomes in patients undergoing high-risk PCI

DETAILED DESCRIPTION:
Although coronary artery bypass grafting is generally preferred in symptomatic patients with severe, complex multivessel, or left main disease, some patients present with clinical features that make coronary artery bypass grafting clinically unattractive. Percutaneous coronary intervention (PCI) with hemodynamic support may be feasible for these high-risk patients. Veno-arterial extracorporeal membrane oxygenation (VA-ECMO) can be used to provide hemodynamic support during high-risk PCI procedures. However, ECMO might increase the rates of severe complications, such as bleeding and limb ischemia. Additionally, some patients might not need the support of ECMO. In this context, investigators propose a standby cannulated ECMO strategy, in which femoral cannulas are inserted and connected to primed circuit, and ECMO is initiated when needed. Therefore, investigators will conduct a prospective randomized clinical trial to compare outcomes between standby cannulated ECMO versus prophylactic ECMO in patients undergoing high-risk PCI. Investigators will randomly assign 176 symptomatic patients with complex 3-vessel disease or unprotected left main coronary artery disease or severely depressed left ventricular function to standby cannulated ECMO group (n=88) or prophylactic ECMO (n=88). The primary end point was the 30-day incidence of major adverse events, including all-cause death, myocardial infraction, any repeat revascularization procedure, stroke, PCI failure, limb ischemia, bleeding, surgical revision and renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Clinicians decide to perform PCI during ECMO support.
2. Age of ≥18
3. Patient presents with a compromised ejection fraction of less than 35% or at risk of hemodynamic deterioration, or intervention on the last patent coronary conduit or an unprotected left main artery, or complex 3-vessel disease (SYNTAX score of ≥33)
4. Informed consent

Exclusion Criteria:

1. Subject in cardiogenic shock(need inotrope, pressor or mechanical support to maintain SBP >90mmHg)
2. Presence of moderate to severe aortic insufficiency
3. Severe peripheral vascular disease
4. creatinine≥4mg/dL
5. Liver dysfunction with elevation of liver enzymes and bilirubin levels to ≥ 3x ULN
6. History of recent (within 1 month) stroke or TIA
7. Abnormal coagulation(defined as platelet count ≤50000/mm3 or Fibrinogen ≤1.50g/L)
8. Allergy or intolerance to heparin, aspirin, ADP receptor inhibitors, or documented heparin induced thrombocytopenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Composite rate of 9 major adverse events | 30 days
  included all-cause death, myocardial infraction, repeat revascularization procedure, stroke, percutaneous coronary intervention failure, limb ischemia, bleeding, surgical revision and renal replacement therapy

SECONDARY OUTCOMES:
Platelet drop | 30 days
  Decrease in PLT during hospitalization
Hemoglobin drop | 30 days
  Decrease in Hb during hospitalization
RBC transfusion rate | 30 days
Serum interleukin-6 concentration | 30 days
  Highest level of IL-6 during concentration
Duration of ECMO support | 30 days
  Time on ECMO support
Length of hospital stay | 30 days
  Time of hospitalization
Hospitalization cost | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Xiaotong Hou, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No